CLINICAL TRIAL: NCT05444244
Title: Novel Approaches to Identifying and Engaging Disadvantaged Patients With Alzheimer's Disease (AD) in Clinical Research
Brief Title: A Relational Research Recruitment and Engagement Intervention for Cognitive Aging Research
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 2019-1148; 5K76AG060005 (NIH); A534100 (Other: UW Madison); Emergency Medicine (Other: UW Madison); Protocol Version (Other: UW Madison)
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Results first posted 2024-02-01 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-01

CONDITIONS: Dementia; Cognitive Dysfunction; Alzheimer Disease; Lewy Body Disease; Frontotemporal Dementia
Keywords: Recruitment Intervention; Recruitment Science; Alzheimer's Disease Research Participation
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Alzheimer Disease; Lewy Body Disease; Frontotemporal Dementia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brain Health Community Registry Recruitment (Active Comparator)
  Interventions: Other: Relational Research Recruitment and Engagement Intervention
- Standard Recruitment (No Intervention)

INTERVENTIONS:
Other: Relational Research Recruitment and Engagement Intervention — * Specified recruiter/point of contact
  * Flexibility in study time, place, method of recruitment (preferred participant email, phone), and follow-up (in registry, if participant calls back at all restart 3 failed phone contacts)
  * Resource matching (financial, transportation constraints)
  Other Names: Brain Health Community Registry Recruitment Intervention
  Arms: Brain Health Community Registry Recruitment

SUMMARY:
Despite well-documented disparities in Alzheimer's disease and related dementia (AD) prevalence, incidence, treatment, and mortality, individuals from disadvantaged backgrounds (e.g. racial/ethnic minorities and socioeconomically disadvantaged persons) are under-represented in clinical research. Existing research recruitment approaches are rarely designed to accommodate the priorities, concerns, and constraints relevant to participants from diverse backgrounds. To address these gaps, the investigators developed a research recruitment and engagement model, the Participant Oriented Research Engagement Model that centers and prioritizes relational aspects of research engagement, research participant needs, and systematically address socioeconomic determinants (i.e. unmet needs) that may limit accessibility of research. The investigators propose to test the effectiveness of the Brain Health Community (BHC) Registry recruitment and engagement intervention, as compared to standard research recruitment strategies in modifying enrollment rates, participant satisfaction, and engagement. The investigators hypothesize that the BHC Registry will yield greater enrollment rates, higher satisfaction, and better ratings of relational engagement.

DETAILED DESCRIPTION:
Despite well-documented disparities in Alzheimer's disease and related dementia (AD) prevalence, incidence, treatment, and mortality, individuals from disadvantaged backgrounds (e.g. racial/ethnic minorities and socioeconomically disadvantaged persons) are under-represented in clinical research. This poses a major barrier for efforts to better understand how disease risk factors and protective factors influence ADRD progression, and determinants of observed disparities. The National Institute on Aging has highlighted the need for development of an applied recruitment science to advance ADRD research, and enable systematic investigation of ADRD health disparities. Existing research on optimal ADRD research recruitment, engagement, and retention strategies is sparse, and focuses predominantly on individual-level characteristics, many of which may not be modifiable. Much of this research also overlooks the role of structural and social determinants, along with features of the study design in shaping participation decisions. People with ADRD and their caregivers commonly face financial, social, emotional, and logistical (i.e. time scarcity) consequences in relation to dementia, that disproportionately burden disadvantaged populations, yet are overlooked in research recruitment and engagement approaches. Existing research recruitment approaches are rarely designed to accommodate the priorities, concerns, and constraints relevant to participants from diverse backgrounds.

To address these gaps, the investigators developed a research recruitment and engagement model, the Participant Oriented Research Engagement Model that centers and prioritizes relational aspects of research engagement, research participant needs, and systematically address socioeconomic determinants (i.e. unmet needs) that may limit accessibility of research. Core constructs within the model are implemented within an applied research recruitment and engagement intervention, the Brain Health Community (BHC) Registry which applies systematic, tailored, and relational recruitment strategies and standardized connections to resources as an element of the research engagement process. The investigators propose to test the effectiveness of the BHC Registry recruitment and engagement intervention, as compared to standard research recruitment strategies in modifying enrollment rates, participant satisfaction, and engagement. Each approach will be evaluated in a randomized trial to either BHC Registry or Standard Recruitment (SR). The relative benefit of these two approaches will be evaluated in a crossover trial of 60 participants who will be randomized in a 2:1 ratio. The investigators hypothesize that the BHC Registry will yield greater enrollment rates, higher satisfaction, and better ratings of relational engagement. Upon completion of the study, participants who received SR will be invited to participate in the BHC Registry.

Aim 1: To compare the BHC Registry to SR with respect to enrollment factors.

Aim 2: To compare the BHC Registry to SR with respect to participant satisfaction and relational engagement.

Hypothesis A: Tailored and relational recruitment strategies used in BHC Registry will result in higher enrollment, lower rates of refusal, and lower drop-out rates.

Hypothesis B: Tailored and relational recruitment strategies used in BHC Registry will result in higher participant satisfaction ratings.

Hypothesis C: Tailored and relational recruitment strategies used in the BHC Registry will yield better ratings of relational engagement.

Hypothesis D: Tailored and relational recruitment strategies used in BHC Registry will result in more favorable attitudes toward research as assessed by the Clinical Research Involvement Scale (CRIS)

ELIGIBILITY:
Inclusion Criteria for Participants Ages 40 or Older:

* English-speaking
* Interested in learning about research opportunities related to aging, brain health, and caregiving
* If evidence of a lack of decision-making capacity is present, presence and consent from a legally authorized representative (LAR) in addition to assent from the participant with cognitive challenges

Inclusion Criteria for Caregiver Participants Ages 18 or Older:

* English-speaking
* Has had previous or current contact (phone, in-person, coordination of services, etc.) with a person with Alzheimer's disease or related dementia at least monthly and provides unpaid support to the individual which can be health, financial, social, or logistical in nature
* Interested in learning about research opportunities related to aging and brain health, particularly related to care for people living with Alzheimer's disease or related dementia

Exclusion Criteria for Participants Ages 40 or Older:

* Is not interested in learning about research opportunities related to aging and brain health
* Under 40 years of age and/or no ADRD caregiving experience
* Evidence of a lack of decision-making capacity and LAR cannot be found or contacted
* Populations who are completely blind or completely deaf

Exclusion Criteria for Caregiver Participants Ages 18 or Older:

* Frequency of contact with the person with ADRD is or has been less than monthly
* Nature of contact does not involve providing supports for person with ADRD, or caregiver is paid for supports
* Under 18 years of age
* Populations who are completely blind or completely deaf

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea L Gilmore-Bykovskyi, PhD, RN, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants have been enrolled into the Standard Recruitment arm as of grant closeout on 5/31/2023.
Groups:
- Standard Recruitment: No specified recruiter/point of contact Limited flexibility in study time, place, method of recruitment and follow-up No resource matching
Period: Overall Study
Arm/Group | Brain Health Community Registry Recruitment | Standard Recruitment
Started | 182 | 0 (No participants recruited for this arm as of grant closeout.)
Completed | 182 | 0 (No participants recruited for this arm as of grant closeout.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were recruited for the standard recruitment arm as of study closeout on 5/31/2023.
Groups:
- Standard Recruitment: * No specified recruiter/point of contact
  * Limited flexibility in study time, place, method of recruitment, and follow-up
  * No resource matching
- Total: Total of all reporting groups
Arm/Group | Brain Health Community Registry Recruitment | Standard Recruitment | Total
Number analyzed (Participants) | 182 | 0 | 182
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 72 |  | 72
  >=65 years | 110 |  | 110
Age, Continuous [Mean (Full Range); unit: years] | 65.87 [36 to 99] |  | 65.87 [36 to 99]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 |  | 134
  Male | 48 |  | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 |  | 2
  Asian | 1 |  | 1
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 2 |  | 2
  White | 171 |  | 171
  More than one race | 6 |  | 6
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 182 |  | 182
Participants Requesting Resources [Count of Participants; unit: Participants] | 97 |  | 97

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Enrolled in Each Recruitment Arm
Description: Number of participants enrolled in the Brain Health Community Registry
Time Frame: 10 months
Population: No participants were enrolled in the Standard Recruitment arm as of study closeout (5/31/2023). Analysis only accounts for the Brain Health Community Registry Recruitment Arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Brain Health Community Registry Recruitment | Standard Recruitment
Number analyzed (Participants) | 182 | 0
Participants | 182 |

2. Secondary Outcome: Number of Participants Retained Over Time
Description: Number of participants in the Brain Health Community Registry
Time Frame: 10 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Brain Health Community Registry Recruitment | Standard Recruitment
Number analyzed (Participants) | 182 | 0
Participants | 182 |

3. Other Pre Specified Outcome: Participants Matched With Resources
Description: As part of the Brain Health Community Registry, participants were given the option to have a tailored list of resources created for them. Resources included transportation needs, caregiving support groups, resources related to eyeglasses or hearing aids, food, and other needs. This measure indicates the number of participants out of the 182 total participants that requested and received a personal resource list.
Time Frame: 10 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Brain Health Community Registry Recruitment: Relational Research Recruitment and Engagement Intervention: • Specified recruiter/point of contact
  * Flexibility in study time, place, method of recruitment (preferred participant email, phone), and follow-up (in registry, if participant calls back at all restart 3 failed phone contacts)
  * Resource matching (financial, transportation constraints)
Arm/Group | Brain Health Community Registry Recruitment | Standard Recruitment
Number analyzed (Participants) | 182 | 0
Participants | 97 |

ADVERSE EVENTS:
Time Frame: 10 months
Description: No participants were enrolled in the Standard Recruitment arm as of study closeout (5/31/2023). Risk for Serious Adverse Events, All-Cause Mortality, and Other (Not Including Serious) Adverse Events only accounts for the Brain Health Community Registry Recruitment Arm.
Arm/Group | Brain Health Community Registry Recruitment | Standard Recruitment
All-Cause Mortality (participants affected / at risk) | 0/182 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/182 | 0/0
Other Adverse Events (participants affected / at risk) | 0/182 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-31): https://cdn.clinicaltrials.gov/large-docs/44/NCT05444244/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-07): https://cdn.clinicaltrials.gov/large-docs/44/NCT05444244/ICF_001.pdf